CLINICAL TRIAL: NCT02359487
Title: Behavioral Counseling Intervention Trial to Reduce Alcohol-related Sexual Risk Behavior Among HIV-negative Men in Namibia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6031
Record Dates: First submitted 2015-01-28; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Alcohol Consumption; Alcohol Abuse; HIV; Sexual Behavior
Keywords: Namibia; Alcohol; HIV; Sexual risk
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Sexual Behavior | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention consists of a 1-hour individual counseling session relating to alcohol consumption and HIV sexual risk behaviors. Intervention counselors will assess alcohol-related sexual risk behaviors through the use of job aids that include a flip chart, guided scripts, activities, role plays, and a take home booklet. Counselors use motivational interviewing and interactive activities to discuss alcohol and HIV myths and facts, participants personal risk behaviors, and a decision-making activity that assists participants in weighing the pros and cons of engaging in risky behavior. Counselors also facilitate role plays to improve communication skills in risky situations, as well as a condom demonstration and skills session, and goal setting. In addition, men in the intervention arm will also receive two cell phone text messages 1-month and 4-months following enrollment to reiterate risk reduction messages.
  Interventions: Behavioral: Alcohol-HIV Risk Reduction Counseling
- Control (Placebo Comparator): Participants assigned to the control arm will be given a general alcohol information booklet and an alcohol abuse support services brochure. The alcohol information booklet contains information about responsible drinking, signs and symptoms of alcohol abuse, advice and guidance to reduce alcohol intake, and resources for assistance. The alcohol support services brochure contains times, dates, and locations of peer support and counseling services in the Windhoek region.
  Interventions: Behavioral: Placebo Intervention

INTERVENTIONS:
Behavioral: Alcohol-HIV Risk Reduction Counseling — The intervention consists of a 1-hour individual counseling session relating to alcohol consumption and HIV sexual risk behaviors. Intervention counselors will assess alcohol-related sexual risk behaviors through the use of job aids that include a flip chart, guided scripts, activities, role plays, and a take home booklet. Counselors use motivational interviewing and interactive activities to discuss alcohol and HIV myths and facts, participants personal risk behaviors, and a decision-making activity that assists participants in weighing the pros and cons of engaging in risky behavior. Counselors also facilitate role plays to improve communication skills in risky situations, as well as a condom demonstration and skills session, and goal setting. In addition, men in the intervention arm will also receive two cell phone text messages 1-month and 4-months following enrollment to reiterate risk reduction messages.
  Arms: Intervention
Behavioral: Placebo Intervention — Participants assigned to the control arm will be given a general alcohol information booklet and an alcohol abuse support services brochure. The alcohol information booklet contains information about responsible drinking, signs and symptoms of alcohol abuse, advice and guidance to reduce alcohol intake, and resources for assistance. The alcohol support services brochure contains times, dates, and locations of peer support and counseling services in the Windhoek region.
  Arms: Control

SUMMARY:
The overall purpose of this study is to evaluate an intervention that aims to reduce alcohol-related HIV sexual risk behaviors among HIV-negative men in Namibia. The objectives of the study are to determine the effectiveness of an individual counseling intervention in reducing alcohol-related HIV sexual risk behaviors among men, and in reducing harmful and hazardous alcohol use among men.

DETAILED DESCRIPTION:
This study involves a randomized controlled trial of 550 HIV-negative adult men recruited from a single Voluntary Counseling and Testing (VCT) center for HIV in Windhoek, Namibia who report harmful or hazardous alcohol consumption and more than one sex partner in the previous three months.

After receiving standard counseling at the VCT center, all men who test HIV-negative will be invited to be screened for eligibility for the study, and if eligible, to consent to enroll. Personnel hired for the study will then administer a baseline survey via Personal Digital Assistant to all enrolled men. Enrolled participants will then be randomized to either an intervention arm, and receive an additional one-hour counseling session and take-home materials plus general alcohol information materials or to a control arm, and receive general alcohol information materials alone. All men enrolled in the study will receive the general alcohol information materials, consisting of a booklet with alcohol health information and a brochure detailing alcohol abuse support services in the local community. Men in the intervention arm will also receive two cellphone text messages one month and four months following enrollment to boost the risk reduction counseling. Follow-up surveys of all participants will be conducted three months and six months after enrollment

Outcomes measured include self-reported data at baseline, three months and six months post-enrollment regarding: 1) Number, proportion of sex acts preceded by alcohol use; 2) Number, proportion of sex acts protected by condoms; 3) Number of sex partners; and 4) Quantity and frequency of alcohol use; 5) Condom use demonstration scores.

ELIGIBILITY:
Inclusion Criteria:

* Self reported HIV negative status after testing at the Council of Churches Namibia (CCN) NewStart VCT center
* More than 1 sexual partner in the past 6 months
* AUDIT screen score 8 to 19
* Able to provide informed consent
* Access to a cell phone to retrieve private text messages and calls
* Plans to stay in the local area for 6 months
* Able to verbally communicate in English, Oshiwambo, or Afrikaans

Exclusion Criteria:

* Self reported HIV positive status after testing at the CCN NewStart VCT center
* Less than 1 sexual partner in the past 6 months
* AUDIT screen score less than 8 or greater than 20
* Unable to provide informed consent to participate to enroll in the study
* Unable to retrieve private cell phone text messages and calls
* Unable to verbally communicate in English, Oshiwambo, or Afrikaans

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in frequency of sex after drinking (measured by count data and proportions) | 3 months, 6 months after intervention
  Sex acts preceded by alcohol use, for up to 4 recent sex partners, measured by count data and proportions

SECONDARY OUTCOMES:
Change in frequency of condom use (measured by count data and proportions) | 3 months, 6 months after intervention
  Sex acts protected by condoms, for up to 4 recent sex partners, measured by count data and proportions
Change in number of sex partners | 3 months, 6 months after intervention
  Number of sex partners in preceding 6 months
Change in frequency of alcohol use (measured by AUDIT and CAGE screens) | 3 months, 6 months after intervention
  Quantity and frequency of alcohol use, measured by AUDIT and CAGE screens
Change in condom skills (measured by a condom use demonstration score, modified 9-item male condom use score (MCUS) | 3 months, 6 months after intervention
  Changes in condom skills, as measured by a condom use demonstration score

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Bock, MD, Principal Investigator — Centers for Disease Control and Prevention